CLINICAL TRIAL: NCT01021631
Title: Transfusion Requirements After Cardiac Surgery: a Randomized Controlled Clinical Trial (TRACS STUDY)
Brief Title: TRACS STUDY: Transfusion Requirements After Cardiac Surgery
Acronym: TRACS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Jose Otavio Costa Auler Jr, InCor - HCFMUSP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Transfusion
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery; Strategies of transfusion; Red blood cells; Liberal; Restrictive; Anemia
MeSH Terms: conditions — Anemia | interventions — Erythrocyte Transfusion; Erythrocyte Count; Blood Transfusion; Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal Transfusion Strategy (Active Comparator): Liberal Group - transfusion when hematocrit is lower than 30%
  Interventions: Other: Red blood cell transfusion
- Restrictive Transfusion Strategy (Active Comparator): Restrictive Group - transfusion when hematocrit is lower than 24%
  Interventions: Other: Red blood cell transfusion

INTERVENTIONS:
Other: Red blood cell transfusion — Red blood cell (RBC) transfusion will be given when hematocrit fall below 30% since intraoperative until the discharge of intensive care unit. Following administration of the 1 RBC unit, a repeat hematocrit is performed;if a patient's hematocrit is 30% or higher, no additional transfusion is necessary.
  Other Names: Red blood cells; Transfusion; Liberal; Cardiac surgery
  Arms: Liberal Transfusion Strategy
Other: Red blood cell transfusion — Red blood cell (RBC) transfusion will be only given when hematocrit fall below 24% since intraoperative until the discharge of intensive care unit. Following administration of the 1 RBC unit, a repeat hematocrit is performed;if a patient's hematocrit is 24% or higher, no additional transfusion is necessary.
  Other Names: Red blood cells; Transfusion; Restrictive; Cardiac surgery
  Arms: Restrictive Transfusion Strategy

SUMMARY:
Blood transfusion is related to worse outcomes and the triggers for red blood cells transfusion are not well defined in cardiac surgery. Retrospective studies in cardiac surgery do not show benefits of red blood cell transfusion in reduction of morbidity and mortality in cardiac surgery. There are no prospective studies comparing outcomes between restrictive or liberal strategy in cardiac surgery.This study is a double-blind randomized study comparing clinical outcomes between two strategies of transfusion in cardiac surgery - liberal or restrictive.

DETAILED DESCRIPTION:
Blood transfusion is commonly performed in patients submitted to cardiac surgery. However, there are many studies reporting adverse effects of this intervention and final data on benefits are not available. There are no prospective studies in cardiac surgery regarding red blood cell transfusions requirements. There are retrospective studies in cardiac surgery suggesting worse outcomes including higher rates of mortality in patients submitted to red blood transfusion. Hematocrit levels around 30% are usually recommended not evidence based. Our purpose is to prospectively evaluate two strategies of transfusion in 500 patients submitted to elective cardiac surgery: a liberal strategy - patients receive blood transfusion when hematocrit is lower than 30% since the intraoperative period until the ICU discharge; a restrictive strategy - patients receive blood transfusion only when hematocrit is lower than 24%.

Clinical outcomes, costs and quality of life will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All elective primary and redo adult cardiac surgical patients for coronary artery bypass grafting, valve procedure or combined procedures
* Adults patients
* Written informed consent

Exclusion Criteria:

* Age less than 18 years
* Transplant procedures
* Emergency procedures
* Aortic repairs
* Congenital procedures
* Previous anemia (hemoglobin lower than 10 g/dL)
* Previous thrombocytopenia (platelet number lower than 100.000/mm3)
* Previous known coagulopathy
* Pregnancy
* Those unable to receive blood transfusion
* Patients who refused participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The primary purpose of this study is to compare clinical outcomes after cardiac surgery in patients submitted to different strategies of red blood cell transfusion | 30 days after surgery

SECONDARY OUTCOMES:
To compare length of stay in ICU, length of stay in Hospital, health-related quality of life, hospital costs and mortality between groups. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila A Hajjar, MD, Principal Investigator — InCor - HCFMUSP
Locations (1):
- InCor - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Hajjar LA, Auler Junior JO, Santos L, Galas F. Blood tranfusion in critically ill patients: state of the art. Clinics (Sao Paulo). 2007 Aug;62(4):507-24. doi: 10.1590/s1807-59322007000400019. PMID 17823715
- [Background] Auler JO Jr, Galas F, Hajjar L, Santos L, Carvalho T, Michard F. Online monitoring of pulse pressure variation to guide fluid therapy after cardiac surgery. Anesth Analg. 2008 Apr;106(4):1201-6, table of contents. doi: 10.1213/01.ane.0000287664.03547.c6. PMID 18349193
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Nakamura RE, Vincent JL, Fukushima JT, de Almeida JP, Franco RA, Lee Park C, Osawa EA, Pinto Silva CM, Costa Auler JO Jr, Landoni G, Barbosa Gomes Galas FR, Filho RK, Hajjar LA. A liberal strategy of red blood cell transfusion reduces cardiogenic shock in elderly patients undergoing cardiac surgery. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1314-20. doi: 10.1016/j.jtcvs.2015.07.051. Epub 2015 Jul 26. PMID 26318355
- [Derived] Galas FR, Almeida JP, Fukushima JT, Osawa EA, Nakamura RE, Silva CM, de Almeida EP, Auler JO, Vincent JL, Hajjar LA. Blood transfusion in cardiac surgery is a risk factor for increased hospital length of stay in adult patients. J Cardiothorac Surg. 2013 Mar 26;8:54. doi: 10.1186/1749-8090-8-54. PMID 23531208
- [Derived] Hajjar LA, Almeida JP, Fukushima JT, Rhodes A, Vincent JL, Osawa EA, Galas FR. High lactate levels are predictors of major complications after cardiac surgery. J Thorac Cardiovasc Surg. 2013 Aug;146(2):455-60. doi: 10.1016/j.jtcvs.2013.02.003. Epub 2013 Mar 15. PMID 23507124
- [Derived] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381